CLINICAL TRIAL: NCT05111899
Title: Leading Advancements in the Uptake of Newborn Community Health (LAUNCH)
Brief Title: Leading Advancements in the Uptake of Newborn Community Health
Acronym: LAUNCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Frankel Family Foundation (Unknown); Stewardship Foundation (Unknown)
Responsible Party: Principal Investigator, Brandon Guthrie, Associate Professor, School of Public Health: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006942
Record Dates: First submitted 2021-07-26; First posted 2021-11-08 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Breastfeeding, Exclusive; Immunization; Infection; Growth; Stunting, Nutritional
Keywords: Community health worker
MeSH Terms: conditions — Breast Feeding; Infections; Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Newborn Health Education
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Newborn Health Education — Community influencers will receive training and give community education to women and their families regarding newborn health.
  Arms: Intervention

SUMMARY:
The primary objective of the study is to determine the impact of a behavior change intervention that partners Orthodox priests with members of the Health Development Army (HDA) and train them to conduct newborn health outreach to increase rates of early initiation of and exclusive breastfeeding through 6 months and vaccination coverage at six months.

Secondary objectives include:

* Determine the impact of the intervention on infant growth at six months, observed and self-reported changes in nutrition and feeding practices of mother and infants, and early identification of newborn illness.
* Design a culturally relevant, scalable intervention for community-based newborn and infant health in Gondar in partnership with local partners, the Federal Ministry of Health, and the Gondar Regional Health Bureau.

DETAILED DESCRIPTION:
The study will test a model the leverages existing community networks to improve the health of newborns in Gondar, Ethiopia. The intervention will be implemented at the community level by pairs of trained Ethiopian Orthodox priests and members of the Heath Development Army (HDA). A list of priests serving at the EOC churches in the intervention arm will be obtained through the woreda diocese and their respective churches. All the priests will be contacted through the church leadership and asked to participate in the study intervention. The intervention will be implemented in collaboration with HDA members recruited by HEWs under the health centers in the catchment areas of the intervention churches.

An initial 5 day training will be given to priests and HDA members. The training will focus on newborn health topics including early initiation of and exclusive breastfeeding, maternal nutrition, immunization, childhood illnesses, child health care services, etc. At the end of the training action plans will be prepared by the training organizers, priests, and HDA. Priest will be asked to integrate health messages and education into their routine family visits around the birth of a child in structured intervals as culturally appropriate.

The trained priests and HDA members will be dispatched to their respective communities to begin the intervention. Their primary activities will be identification of near-term pregnant and newly delivered women, providing health education to their families, follow-up visits to enable newborn-mother pairs to access child health care services, and to provide health education at religious and community gatherings. Specifically, pre-planned visits of parishioners' families will be done by the respective priests and the partnering HDA members during the last month of pregnancy, immediately after the delivery of the baby and around the time of baptism for the newborn. These visits will be used to educate pregnant and postpartum women and their families on newborn health topics including initiation of breastfeeding, duration of breastfeeding/ exclusive breastfeeding, vaccination, cord care, and utilization of available newborn health care services. These community based activities will be monitored through regular follow-up visits by the UoG study team and discussions with priests and HDA members.

Newborn-mother pairs will be recruited within the first 10 days after delivery as reported to the study team by Health Extension Workers (HEWs) engaged in the study. Recruitment will start one month following the start of the intervention and all reported newborn-mother pairs who meet the screening criteria will be included in the study until the calculated sample sizes are reached. HEW's routine registers of new deliveries will be used to trace, recruit and screen study participants. Newborn-mother pairs who fulfill an initial screening criteria will be reported to the study team at the University of Gondar (UoG) who will travel to the study site regularly for recruitment of study participants and data collection. Newborn-mother pairs will be reported to the UoG study team both through phone calls made by HEWs and in-person at the time of regular onsite visits by the team.

Newborn-mother pairs will be recruited within the first 10 days after delivery as reported to the study team by Health Extension Workers (HEWs) engaged in the study. Recruitment will start one month following the start of the intervention and all reported newborn-mother pairs who meet the screening criteria will be included in the study until the calculated sample sizes are reached. HEW's routine registers of new deliveries will be used to trace, recruit and screen study participants. Newborn-mother pairs who fulfill an initial screening criteria will be reported to the study team at the University of Gondar (UoG) who will travel to the study site regularly for recruitment of study participants and data collection. Newborn-mother pairs will be reported to the UoG study team both through phone calls made by HEWs and in-person at the time of regular onsite visits by the team.

Eligible newborn-mother pairs will be visited by a member of the study team at their home or at an appointed meeting location in their community to complete the verbal informed consent process. Those pairs who attend church at a parish that received the intervention will be assigned to the intervention arm, and those from the parishes where no intervention was conducted will be assigned to the control arm. Initial baseline data will then be collected and follow-up visit schedules arranged with the study team.

ELIGIBILITY:
Inclusion Criteria:

Newborn-mother pairs visited by the study staff (Enrolled women and newborns)

The following inclusion criteria will be used during recruitment:

* Newborns should be those delivered at least one month after the start of the intervention period
* Newborn-mother pairs should be EOC parishioners
* Newborn's family should have a soul father (a spiritual advisor assigned to the family in the Ethiopian Orthodox tradition)
* Mother must have lived in the study area for at least 6 months
* Mothers must give written informed consent for themselves and their newborn

Formative focus group discussion and key informant interview participants (FGD and KII participants)

The following inclusion criteria will be used during recruitment:

* Mothers of newborns <6 months old
* Fathers of newborn children <6 months
* Ethiopian Orthodox priests from the North Gondar region
* Healthcare workers from government Health Centers (unit of primary care)
* All participants must have established residency in the region for >6 months
* All participant must give verbal informed consent

Exclusion Criteria:

Newborn-mother pairs visited by the study staff (Enrolled women and newborns)

The following exclusion criteria will be used during recruitment:

* Newborns with gross developmental abnormalities that would make anthropometric measurements and interpretations difficult
* Newborns identified by the study team as in distress and in need of immediate, emergency care during the enrollment visit
* Newborn whose mother is not a member of an EOC parish
* Newborns whose mothers have died by the time of recruitment
* Newborn whose family plans to re-locate away from the study site in less than 6 months
* Newborns who were part of a multiple birth but are not the first born should be excluded

Formative focus group discussion and key informant interview participants (FGD and KII participants)

The following exclusion criteria will be used during recruitment:

- Newly established residence in the Woreda (<6 months)

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 316 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Mid-upper arm circumference | Up to six months
  Anthropometric Measurement using MUAC tapes
Proportion of mothers exclusive breastfeeding | Up to six months
  Self-reported breastfeeding behavior

SECONDARY OUTCOMES:
Immunization status | Up to six months
  Collected from vaccination cards
Frequency of acute illness | Up to six months
  Self reported
Frequency of hospitalization status | Up to six months
  Self reported

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Guthrie, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Gondar, Gonder, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alemie GA, Walson J, Rankin KC, Wild LM, Tesema GA, Belay DG, Hakizimana D, Guthrie BL. Newborn community health advancements among Ethiopian Orthodox Christian women in North Gondar, Ethiopia: community-based randomised trial protocol. BMJ Open. 2024 Sep 13;14(9):e081330. doi: 10.1136/bmjopen-2023-081330. PMID 39277203

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT05111899/Prot_SAP_000.pdf